CLINICAL TRIAL: NCT01855594
Title: Double Blind, Randomized Placebo-controlled Clinical Study Evaluating the Efficacy of Lithium Carbonate in the Treatment of Neuropathic Pain of Patients With Spinal Cord Injury
Brief Title: Study to Evaluate the Efficacy of Lithium Carbonate in Spinal Cord Injury Patients With Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: China Rehabilitation Research Center (Other Government); Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN302
Record Dates: First submitted 2013-05-12; First posted 2013-05-16 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Neuropathic Pain; Neuralgia; Spinal Cord Injuries
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium treatment group (Experimental): Lithium carbonate, 250mg/tablet. The dose starts with three times a day and one tablet each time for a week. The daily dose will then be adjusted according to serum lithium level and clinical finding. Target serum lithium level is 0.6 - 1.2mmol/L.
  Interventions: Drug: Lithium Carbonate
- Control group (Placebo Comparator): The dose of the placebo will be adjusted according to the dummy serum level report.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — 250 mg/tablet, 6 weeks course of oral administration
  Arms: Lithium treatment group
Drug: Placebo — placebo tablet, 6 week course of oral administration
  Arms: Control group

SUMMARY:
To investigate the efficacy of lithium carbonate in the treatment of neuropathic pain of patients with spinal cord injury.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded trial. Sixty spinal cord injured subjects with neuropathic pain will be randomized into two groups. The subject in the Treatment Group will receive lithium carbonate tablet, while the Control Group will receive placebo tablet. Neither the subjects nor the physicians know which group the subjects are allocated.

Each subject will receive 6 weeks of oral lithium carbonate or placebo. In the Treatment Group, the dose will be adjusted according to the serum lithium level. While in the Control Group, the dose will be adjusted based on the dummy serum level report.

The outcome will be assessed during visits at 1 week, 2 weeks, 6 weeks and 12 weeks, and a phone call follow-up at 24 weeks from the start of the medication. The primary outcome measure is the severity level of pain. The efficacy and safety will be analyzed by comparing the results of the Treatment Group with those of the Control Group

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65;
* Diagnosis of traumatic spinal cord injury;
* Clinically diagnosed neuropathic pain;
* Pain severity is at least 4 on a 11-point numeric rating scale at screening;
* Pain present regularly for at least 6 weeks before enrollment;
* Able to understand instructions and provide reliable pain assessments;
* Subjects who are voluntarily signed and dated an Ethics Committee approved informed consent form;

Exclusion Criteria:

* Significant renal, cardiovascular, hepatic, infectious or psychiatric disease;
* Significant brain injury with neurological deficits;
* Debilitation or dehydration;
* Addison's disease;
* Recent (within 1 week) or current use of anti-diuretics or other drugs that interacts with lithium, such as tricyclic antidepressants, nonsteroidal antiinflammatory drug and tetracyclines;
* A history of substance or alcohol abuse within past 1 year;
* A need for elective surgery involving preoperative or postoperative analgesics or anesthetics during the study period;
* Current pregnant or breast feeding, or female who has childbearing potential but is not willing to use an approved method of birth control;
* Participation in any drug study in the last three months;
* History of oral lithium intake for any reason; or
* any criteria, which in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Numeric Rating Scale (NRS) at 24 weeks | D0, Wk 1, 2, 6, 12, and 24
  pain severity level

SECONDARY OUTCOMES:
Change in Multidimensional Pain Inventory Life Interference Subscale (MPI-LIS) | D0, Wk 1, 2, 6, 12 and 24
Change in Short-Form 36 single question | D0, Wk 1, 2, 6, 12, and 24
Change in Sleep Interference Assessment score | D0, Wk 1, 2, 6, 12 and 24
Change in weekly number of days with pain attack | D0, Wk 1, 2, 6, 12 and 24
Change in the Patient Global Impression of Change (PGIC) | Wk 1, 2, 6, and 12
Change in Patient Health Questionnaire (PHQ-9) | D0, Wk 1, 2, 6 and 12
Change in sensory score, motor score and ASIA impairment (AIS) scale | D0, Wk 6 and 12
Change in Modified Ashworth Scale | D0, Wk 6 and 12
Magnetic resonance diffusion tensor imaging (optional) | D0, Wk 6 and 12
Electrophysiology (optional) | D0, Wk 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Xijing He, M.D., Principal Investigator — Xi'an Jiaotong University Second Affiliated Hospital; Jianjun Li, M.D., Principal Investigator — China Rehabilitaition Research Center
Locations (2):
- China (2):
  - Xi'an Jiaotong University Second Affiliated Hospital, Xi’an, Shanxi
  - China Rehabilitation Research Center, Beijing

REFERENCES:
- [Background] Yang ML, Li JJ, So KF, Chen JY, Cheng WS, Wu J, Wang ZM, Gao F, Young W. Efficacy and safety of lithium carbonate treatment of chronic spinal cord injuries: a double-blind, randomized, placebo-controlled clinical trial. Spinal Cord. 2012 Feb;50(2):141-6. doi: 10.1038/sc.2011.126. Epub 2011 Nov 22. PMID 22105463
- [Background] Wong YW, Tam S, So KF, Chen JY, Cheng WS, Luk KD, Tang SW, Young W. A three-month, open-label, single-arm trial evaluating the safety and pharmacokinetics of oral lithium in patients with chronic spinal cord injury. Spinal Cord. 2011 Jan;49(1):94-8. doi: 10.1038/sc.2010.69. Epub 2010 Jun 8. PMID 20531359